CLINICAL TRIAL: NCT05447455
Title: the Efficacy of Transversus Abdominis Plane Block for Analgesia in Comparison With Local Anesthetic Wound Infiltration Post-cesarean Section: A Randomized Comparative Double-blinded Clinical Trial
Brief Title: TAP Block vs LAWI for Analgesia Post-cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN2022
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Obstetric Pain; Obstetric Anesthesia Problems
Keywords: transversus abdominis plane. VAS; visual analogue score; wound infiltration; cesarean section; postoperative pain; analgesia
MeSH Terms: conditions — Labor Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block group (Active Comparator): A 22-gauge spinal needle was introduced from medial to lateral in-plane to the ultrasound probe, and 20 mL of bupivacaine 0.25% was injected under visualization in the plane between the transversus abdominis muscle and the fascia deep to the internal oblique muscle on each side.
  Interventions: Procedure: Transversus Abdominis Plane Block
- LAWI group (Active Comparator): 40 mL of bupivacaine 0.25% was injected subcutaneously into the surgical wound (20 mL on each of the upper and lower sides) by the obstetrician before skin closure
  Interventions: Procedure: Local anesthetic wound infiltration

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — A 22-gauge spinal needle was introduced from medial to lateral in-plane to the ultrasound probe, and 20 mL of bupivacaine 0.25% was injected under visualization in the plane between the transversus abdominis muscle and the fascia deep to the internal oblique muscle on each side.
  Arms: TAP block group
Procedure: Local anesthetic wound infiltration — 40 mL of bupivacaine 0.25% was injected subcutaneously into the surgical wound (20 mL on each of the upper and lower sides) by the obstetrician before skin closure
  Arms: LAWI group

SUMMARY:
Adequate pain control after cesarean delivery is a significant concern both for parturients and obstetric anesthesiologists. Transversus Abdominis Plane (TAP) block and local Wound infiltration with anesthetics are alternatives for reducing the severity of pain, total analgesic consumption, and opioid side effects. Both the TAP block and wound infiltration are superior to placebo; however, it is unknown which provides better analgesia after cesarean delivery because of a scarcity of randomized clinical trials. So, we hypothesized that the TAP block would decrease postoperative pain and postoperative cumulative opioid consumption at 24 hours

ELIGIBILITY:
Inclusion Criteria:

1. Women who underwent cesarean section under spinal anesthesia.
2. Aged ≥19 years and less than 40 years.
3. Gestational age ≥ 37 Weeks.

Exclusion Criteria:

1. Body mass index (BMI) ≥40 kg/m2.
2. History of recent opioid exposure
3. Hypersensitivity to any of the drugs used in the study.
4. Significant cardiovascular, renal, or hepatic disease

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
degree of pain at rest and on movement (hip flexion and coughing) at 2, 4, 6, 12, and 24 hours postoperatively | 24 hours
  , using a visual analog scale (VAS) score for pain intensity reported on 0-10-point scale for analysis. (0 = no pain and 10 = the worst possible pain).

SECONDARY OUTCOMES:
measures the time to the first postoperative opioid dose | 24 hours
cumulative opioid consumption at 2, 4, 6, and 12 hours. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Taymour, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine - Cairo university, Cairo, Kasr El Ainy, Egypt

IPD SHARING:
Plan to Share IPD: Undecided